CLINICAL TRIAL: NCT05932576
Title: A Multicenter Cohort Study Assessing the Efficacy and Adverse Effects of Different HPV Vaccination in Chinese Women
Brief Title: A Multicenter Cohort Study Assessing the Efficacy and Adverse Effects of HPV Vaccination in Chinese Women
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fujian Maternity and Child Health Hospital (Other)
Responsible Party: Principal Investigator, Binhua Dong, Laboratory of Gynecologic Oncology, Fujian Maternity and Child Health Hospital
Other Study IDs: HVAC2302
Record Dates: First submitted 2023-06-28; First posted 2023-07-06 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-06

CONDITIONS: Human Papillomavirus Vaccines; Efficacy, Self; Adverse Effect; China; Woman

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peripheral blood sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The HPV vaccine group: Women aged 9-45 years who received the last dose of HPV vaccine within the past 12 months were included, and each subject was evaluated within 3-12 months after the last dose of HPV vaccine. Adverse reaction symptoms were queried by telephone follow-up and face-to-face, and peripheral blood tube (3ml) was collected to detect the concentration of comprehensive antibody to HPV vaccine.

SUMMARY:
Human papillomavirus (HPV) is currently one of the most common sexually transmitted infections, according to its carcinogenicity is divided into high-risk genotypes and low-risk genotypes, research has confirmed that carcinogenic HPV type continuous infection leads to a higher incidence of condyloma acuminatum and cervical cancer, while increasing the oropharyngeal cancer, vaginal cancer and other related cancer risk. HPV vaccines have been widely introduced worldwide to prevent cancers of the lower genital tract such as cervical, anal and vulvar cancers. For different types of HPV vaccine, divided into domestic bivalent, imported bivalent (GlaxoSmithKline), quadrivalent (Merck) and nine-valent (Merck) HPV vaccine, four vaccines all prevent HPV 16/18 high-risk type infection disease, and the four and nine-valent HPV vaccine prevention genotypes are different, and different price number of protection rates, vaccination objects and immunization procedures are slightly different. At the same time, studies have shown that women after HPV vaccine, arm redness, swelling, heat and pain have a high incidence of adverse reactions, often accompanied by menstrual disorders, sleep problems, emotional irritability, fever, dizziness, headache and other adverse reactions risk, so we plan to design a multicenter cohort study to evaluate the effectiveness of HPV vaccine with different prices. At the same time, the adverse reaction symptoms of HPV vaccine in the female population of appropriate age were monitored.

DETAILED DESCRIPTION:
This study was led by the Fujian Provincial Maternal and Child Health Hospital, with the following research centers: Xiangya Hospital of Central South University, Fujian Provincial Center for Disease Control and Prevention, Shenzhen Maternal and Child Health Hospital, Hubei Provincial Maternal and Child Health Hospital, Shandong Province and Shaanxi Province. Recruitment was conducted in 6 provinces in different regions of China, and 2000 subjects were recruited in each province. A total of 12,000 subjects were recruited. Each subject was evaluated within 3 to 12 months after the last dose of HPV vaccine, and adverse reaction symptoms were queried by telephone follow-up and face-to-face. Peripheral blood 1 tube (3ml) was collected to detect the concentration of comprehensive antibodies to HPV vaccine. A multicenter cohort study was conducted to evaluate the effectiveness of HPV vaccine and to monitor the symptoms of adverse reactions to HPV vaccine in the female population of appropriate age.

ELIGIBILITY:
Inclusion Criteria:

- Female, aged 9-45; Get the last dose of HPV vaccine within 12 months.

Exclusion Criteria:

- Pregnancy or lactation during HPV vaccination; Those who refuse follow-up and informed consent.

Ages: 9 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Women aged 9-45 years who received their last dose of HPV vaccine within 12 months
Sampling Method: Non-Probability Sample
Enrollment: 12000 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
HPV vaccine neutralizing antibody detection | Within 3 to 12 months of each subject's last dose of HPV vaccine
  All participants were tested for neutralizing antibodies to the HPV vaccine

CONTACTS AND LOCATIONS:
Overall Officials: Sun Pengming, PhD, Study Chair — Fujian Maternity and Child Health Hospital, Affiliated Hospital of Fujian Medical University
Locations (5):
- China (5):
  - Fujian Maternity and Child Health Hospital, Fuzhou, Fujian
  - Fujian Provincial Center for Disease Control and Prevention, Fuzhou, Fujian
  - Maternal and Child Health Hospital of Shenzhen Province, Shenzhen, Guangdong
  - Maternal and Child Health Hospital of Hubei Province, Wuhan, Hubei
  - Xiangya Hospital, Central South University, Changsha, Hunan